CLINICAL TRIAL: NCT07217639
Title: Clinical Validation of the Aptitude Medical Systems Metrix Respiratory Panel Test in At-Home/Non-Laboratory Settings
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aptitude Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TP-25-041; 75A50123C00013 (Other Grant/Funding Number: BARDA)
Record Dates: First submitted 2025-10-14; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: COVID -19; Influenza A; Influenza B; Respiratory Synctial Virus; RSV; Rhinovirus
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- OTC Study (Experimental): This OTC study will take place in simulated home environments which will be set up within or near clinical settings (e.g., urgent care facilities). The study will enroll symptomatic subjects only. Candidate samples will be self-collected by participants (or collected by a guardian for participants under the age of 14 years) and comparator samples will be collected by a healthcare practitioner with informed consent and Institutional Review Board (IRB) approval. Each sample will be coded for confidentiality.
  Interventions: Diagnostic Test: Aptitude Medical Systems Respiratory Panel Test

INTERVENTIONS:
Diagnostic Test: Aptitude Medical Systems Respiratory Panel Test — The Metrix Respiratory Panel Test is a real-time reverse transcription loop-mediated isothermal amplification reaction (RT-LAMP) test that has been designed to detect viral RNA from SARS-CoV-2, Influenza A, Influenza B, Respiratory Syncytial Virus, and Rhinovirus via electrochemical detection using the Metrix Reader. Detection of SARS-CoV-2, Influenza A, Influenza B, Respiratory Syncytial Virus, and Rhinovirus gene targets will produce a positive result, differentiated by each target. If no target is detected and the internal control amplifies, the result is negative. If no amplification is detected in any of the channels, an invalid result is displayed.

SUMMARY:
The Metrix Respiratory Panel Test will be evaluated for use in Non-Laboratory settings in a home testing environment utilizing the clinical study design described herein. The study will take place in simulated home environments which will be set up within or near active clinical settings (e.g., urgent care facilities). This will be a prospective study conducted at three or more investigational sites located within the United States for the clinical validation of the Metrix Respiratory Panel Test for the detection of SARS-CoV-2, Influenza A, Influenza B, Respiratory syncytial virus, and Rhinovirus in anterior nares (AN) swab samples. Additional sites may be added to the study in order to meet minimum subject/sample enrollment requirements and geographic prevalence of respiratory virus infections. Comparator testing will be performed to determine the infection status of each sample for comparison to results generated by the candidate test. The primary comparator for the study will be an FDA-cleared assay for the detection of SARS-CoV-2, Influenza A, Influenza B, Respiratory Syncytial Virus, and Rhinovirus.

DETAILED DESCRIPTION:
The Metrix Respiratory Panel Test will be evaluated for OTC use in a home use testing environment utilizing the clinical study design described herein. The study will take place in simulated home environments which will be set up within or near active clinical settings (e.g., urgent care facilities). This will be a prospective study conducted at three or more investigational sites located within the United States for the clinical validation of the Metrix Respiratory Panel Test for the differential detection of SARS-CoV-2, Influenza A, Influenza B, Respiratory syncytial virus, and Rhinovirus in AN swab samples. Additional sites may be added to the study in order to meet minimum subject/sample enrollment requirements and geographic prevalence of respiratory virus infections. Comparator testing will be performed to determine the infection status of each sample for comparison to results generated by the candidate test. The primary comparator for the study will be an FDA-cleared assay for detection of SARS-CoV-2, Influenza A, Influenza B, Respiratory syncytial virus, and Rhinovirus.

The candidate device, Metrix Respiratory Panel Test, will be evaluated with AN swab sample types. Each Metrix Respiratory Panel Test kit contains all supplies needed to test AN swab samples, including a corresponding QRI for detailed instructions.

This OTC study will take place in simulated home environments which will be set up within or near clinical settings (e.g., urgent care facilities). The study will enroll symptomatic subjects only. Candidate samples will be self-collected by participants (or collected by a guardian for participants under the age of 14 years) and comparator samples will be collected by a healthcare practitioner with informed consent and Institutional Review Board (IRB) approval. Each sample will be coded for confidentiality.

For each participant, a comparator NP swab sample will be obtained by a healthcare practitioner after testing with the candidate device. This NP swab will be tested with the FDA-cleared SARS-CoV-2 assay according to the IFU and will serve as the primary comparator for swab samples. An additional AN swab sample will be collected and stored frozen and dry for later analysis to support future research validation studies.

No results from the investigational test or comparator testing will be used for clinical diagnosis, management of study participants, or to make treatment decisions.

Test results from the Metrix Respiratory Panel Test (investigational test) will be compared to the test results generated from the comparator assay.

No investigational test results will be used for any treatment decisions.

This work is supported by funding provided by the Biomedical Advanced Research and Development Authority (BARDA).

ELIGIBILITY:
Inclusion Criteria:

1. Participant or guardian understands and is able and willing to provide written informed consent, and assent where applicable, prior to study enrollment.
2. Participant is currently exhibiting signs/symptoms of respiratory tract infection including but not limited to fever, cough, sore throat, runny nose, myalgia, headache, chills, new loss of taste or smell, or fatigue. Participant must still be exhibiting symptoms on the day of specimen collection. Days post symptom onset is not to exceed 14 days.
3. Participant or guardian agrees to read, and is able to read with understanding, the Quick Reference Instructions (QRI) prior to beginning the execution of each of the tests.
4. Participant or guardian is able and willing to contribute the required swab specimens for testing and understands and is able and willing to sign the study informed consent.
5. Participant is willing to provide all samples and run tests for the specified investigational devices.

Exclusion Criteria:

1. Participant does not understand and/or is not able and willing to sign the study informed consent and/or assent.
2. Participant or guardian is not able to comply with nasal swab collection requirements following the Quick Reference Instructions (QRI).
3. Participant is not currently exhibiting respiratory tract infection symptoms.
4. Participant has previously participated in the study.
5. Participant is not able to tolerate specimen collection.
6. Participant is currently undergoing or has within the past thirty (30) days undergone treatment with prescription medication to treat SARS-CoV-2 infection, including but not limited to Remdesivir (Veklury®), Nirmatrelvir/Ritonavir (Paxlovid®), Molnupiravir (LagevrioTM) or receiving convalescent plasma therapy for SARS-CoV- 2.
7. Participant is currently undergoing or has within the past thirty (30) days undergone an inhaled influenza vaccine (FluMist®), or antiviral treatment, including but not limited to Amantadine (Symmetrel®), Rimantadine (Flumadine®), Zanamivir (Relenza®), Oseltamivir (Tamiflu®), Baloxavir Marboxil (Xofluza®), Amantadine (Symmetrel®), Rimantadine (Flumadine®), or Peramivir (Rapivab®).
8. Participant is currently undergoing or has within the past thirty (30) days undergone antiviral treatment for RSV, including but not limited to Ribavirin (Virazole®), RSV-IGIV (RespiGam®), Palivizumab (Synagis®), or Nirsevimab-alip (Beyfortus®).
9. Participants who have had a nasal wash or aspirate as part of their standard of care treatment on day of study visit prior to the study sample collection.
10. Participants who have had recent craniofacial injury or surgery, including to correct deviation of the nasal septum, within the previous six (6) months.
11. Participants who do not understand/read the English language.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative detection of RNA from SARS-CoV-2, Influenza A, Influenza B, Respiratory Syncytial Virus, and Rhinovirus, and Measurement of Positive/Negative Percent Agreement with FDA-cleared comparator test | 25 minutes
  Qualitative detection of RNA from SARS-CoV-2, Influenza A, Influenza B, Respiratory Syncytial Virus, and Rhinovirus in unprocessed AN swab samples. Primary objective of this study is to evaluate the performance (positive percent agreement, negative percent agreement and 95% confidence intervals for upper and lower bounds) of the Metrix Respiratory Panel Test for the qualitative detection of SARS-CoV-2, Influenza A, Influenza B, Respiratory Syncytial Virus, and Rhinovirus viral RNA using AN swab samples. Comparator testing will be performed to determine the status of each sample for comparison to results produced by the candidate test. Comparator testing will be performed to determine the infection status of each sample for comparison to results generated by the candidate test. The primary comparator for the study will be an FDA-cleared assay that detects SARS-CoV-2, Influenza A, Influenza B, Respiratory Syncytial Virus, and Rhinovirus.

CONTACTS AND LOCATIONS:
Overall Officials: Brad W Killingsworth, M.A., Principal Investigator — Aptitude Medical Systems, Inc
Locations (1):
- AFC Trussville, Trussville, Alabama, United States

IPD SHARING:
Plan to Share IPD: No